CLINICAL TRIAL: NCT04026087
Title: Characterization of the Subclass of Donor-specific Antibody Determined in Mass Spectrometry as a Risk Factor of Antibody Mediated Rejection in Renal Transplantation
Brief Title: Subclass of Donor-specific Antibody as a Risk Factor of Antibody Mediated Rejection in Renal Transplantation
Acronym: COR-HUM
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0455 UF7724
Record Dates: First submitted 2019-07-11; First posted 2019-07-19 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Antibody-mediated Rejection
Keywords: Renal transplantation; antibody-mediated rejection; DSA; mass spectrometry technique

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with kidney transplant: Blood sample will be took from subjects during this research

SUMMARY:
Antibody-mediated rejection is now recognized as the first cause of long-term kidney transplant loss. This type of rejection is mediated by the presence of graft-specific antibodies, usually directed against HLA (Human Leukocyte Antigens), called DSA (Donor Specific Antibody).

De novo DSA (ie, post-transplantation) is detected in approximately 20% of transplant recipients in the first five years, and is a major risk factor for antibody mediated rejection and graft loss.

All anti-HLA antibodies therefore do not have the same pathogenicity. Some teams have shown that the detection of IgG3 anti-HLA by cytometry is associated with a higher risk of humoral rejection but these results have not been confirmed by others. One of the limitations of the cytometry by Luminex technique is that it only informs the detection of each subclass but does not allow analysis of the distribution of the different subclasses of a DSA.

A method has been developed for the relative detection and quantification of different subclasses of the DSA using the mass spectrometry technique and will be tested during this study. This new quantification method therefore opens up the prospect of studying whether, not only the presence but especially the distribution of IgG subclasses, in particular IgG3, could constitute a reliable and robust marker of humoral rejection.

DETAILED DESCRIPTION:
Antibody-mediated rejection is now recognized as the first cause of long-term kidney transplant loss. This type of rejection is mediated by the presence of graft-specific antibodies, usually directed against HLA (Human Leukocyte Antigens), called DSA (Donor Specific Antibody). It results from the interaction between DSA and HLA present on the surface of graft endothelial cells, complement activation, endothelial cell activation and recruitment of inflammatory cells within the renal microcirculation leading to a graft dysfunction.

De novo DSA (ie, post-transplantation) is detected in approximately 20% of transplant recipients in the first five years, and is a major risk factor for antibody mediated rejection and graft loss. However, the presence of a DSA is not always associated with humoral rejection.

All anti-HLA antibodies therefore do not have the same pathogenicity. The antibody titre (assessed by the fluorescence average (MFI) on Luminex beads) is involved in the risk of rejection but is far from explaining the disparities in clinical evolution.

DSA are mainly IgG of different subclasses whose distribution could have a major impact on their pathogenicity. Indeed, complement-dependent cytotoxicity (CDC) and antibody-dependent cellular cytotoxicity (ADCC) functions differ according to IgG subclass. IgG3 is the subclass that has the greatest potential for complement activation followed by IgG1. IgG3 and IgG1 are also the two subclasses with the best affinities for the FcγRIIIa activating receptor for ADCC mediated by Natural Killer (NK) cells.

Some teams have shown that the detection of IgG3 anti-HLA by cytometry is associated with a higher risk of humoral rejection but these results have not been confirmed by others. One of the limitations of the cytometry by Luminex technique is that it only informs the detection of each subclass but does not allow analysis of the distribution of the different subclasses of a DSA.

A method has been developed for the relative detection and quantification of different subclasses of the DSA using the mass spectrometry technique and will be tested during this study. This new quantification method therefore opens up the prospect of studying whether, not only the presence but especially the distribution of IgG subclasses, in particular IgG3, could constitute a reliable and robust marker of humoral rejection.

ELIGIBILITY:
Inclusion Criteria:

* - Patients over 18 years old
* Renal transplant patients followed at the University Hospital of Montpellier presenting a DSA de novo during follow-up.
* Affiliation or beneficiary of a social security scheme.

Inclusion criteria specific to patients whose graft biopsy has already been performed

* Patients who consented to the collection of a plasma sample on graft biopsy day and use in future programs (Collection DC-2014-2328)
* Collection of non-opposition to participate in the study

Inclusion criteria specific to patients whose biopsy of the graft has not already been performed:

* Eligible for graft biopsy for humoral-mediated rejection (according to Banff 2015 classification) (Appendix 1)
* Collection of non-opposition to participate in the study
* Signature of informed consent to participate in the collection of a plasma sample on graft biopsy day and use in future programs (Collection DC-2014-2328)

Exclusion Criteria:

* Pregnant or lactating women according to Article L1121 5 of the health public Code
* Vulnerable persons according to article L1121-6 of the health public Code
* Major persons placed under guardianship or curator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years old and over with kidney transplant and who have DSA
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
distribution of DSA IgG subclasses | day 0 (inclusion visit)
  the performance of the distribution of DSA IgG subclasses for the diagnosis of humoral rejection in renal transplant patients with Donor Specific Antibodies

SECONDARY OUTCOMES:
histological criteria for humoral rejection | day 0 (inclusion visit)
  Link between the distribution of DSA IgG subclasses and histological criteria for humoral rejection (according to the Banff International Classification 2015)
degradation of graft function | 1 year after inclusion of subjects
  Link between the distribution of DSA IgG subclasses and degradation of graft function (glomerular filtration rate loss of more than 25%)
graft loss | 1 year after inclusion of subjects
  Link between the distribution of DSA IgG subclasses and graft loss

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Pernin, Doctor, Principal Investigator — UH Montpellier
Locations (1):
- CHU Lapeyronie, Montpellier, Hérault, France

REFERENCES:
- [Result] Pernin V, Bec N, Beyze A, Bourgeois A, Szwarc I, Champion C, Chauvin A, Rene C, Mourad G, Merville P, Visentin J, Perrochia H, Couzi L, Larroque C, Le Quintrec M. IgG3 donor-specific antibodies with a proinflammatory glycosylation profile may be associated with the risk of antibody-mediated rejection after kidney transplantation. Am J Transplant. 2022 Mar;22(3):865-875. doi: 10.1111/ajt.16904. Epub 2021 Dec 18. PMID 34863025
- [Result] Pernin V, Beyze A, Szwarc I, Bec N, Salsac C, Perez-Garcia E, Mourad G, Merville P, Visentin J, Perrochia H, Larroque C, Couzi L, Le Quintrec M. Distribution of de novo Donor-Specific Antibody Subclasses Quantified by Mass Spectrometry: High IgG3 Proportion Is Associated With Antibody-Mediated Rejection Occurrence and Severity. Front Immunol. 2020 Jun 2;11:919. doi: 10.3389/fimmu.2020.00919. eCollection 2020. PMID 32670261